CLINICAL TRIAL: NCT04570280
Title: Comparison of the Effects of Aerobic and Resistive Exercises on Sonographic Muscle Measurements, Functional Status, Body Composition and Quality of Life in Female Patients With Rheumatoid Arthritis
Brief Title: Comparison of the Effects of Aerobic and Resistive Exercises in Female Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2915
Record Dates: First submitted 2020-09-14; First posted 2020-09-30 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis; Exercise; Exercise Therapy
Keywords: Rheumatoid Arthritis; Exercise Therapy; Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Range of Motion Exercises (Placebo Comparator): The patients in the control group will be given the practice of range of motion exercises for 12 weeks, 3 days a week for 50 minutes (1 day accompanied by a physiotherapist).
  Interventions: Other: Range of Motion Exercises
- Range of Motion and Resistive Exercises Group (Active Comparator): Patients in this group will be given joint range of motion and resistive exercises with sandbag to the lower extremity for 12 weeks, 3 days a week for 50 minutes (1 day in the presence of a physiotherapist). For the exercises with resistance, the repetition maximum will be calculated and the intensity of the exercises will be adjusted in accordance with the DeLorme protocol.
  Interventions: Other: Resistive Exercises; Other: Range of Motion Exercises
- Range of Motion and Aerobic Exercises Group (Active Comparator): Joint range of motion exercises and aerobic exercises on the treadmill will be given to the aerobic exercise arm, 3 days a week for 12 weeks (1 day in the presence of a physiotherapist). For aerobic exercises, the maximum heart rate of the patients will be calculated during exercise and the exercise intensity will be determined by increasing the target heart rate level during the exercise.
  Interventions: Other: Aerobic Exercises; Other: Range of Motion Exercises

INTERVENTIONS:
Other: Aerobic Exercises — Aerobic exercises with treadmill will be applied 3 times a week for 12 weeks.
  Arms: Range of Motion and Aerobic Exercises Group
Other: Resistive Exercises — Resistive exercises with sandbag will be applied 3 times a week for 12 weeks.
  Arms: Range of Motion and Resistive Exercises Group
Other: Range of Motion Exercises — Range of Motion Exercises will be applied 3 times a week for 12 weeks.

SUMMARY:
It is aimed to objectively demonstrate and compare the effectiveness of aerobic and resistant exercises performed on female patients with rheumatoid arthritis with sonographic muscle measurements. In addition, it is planned to compare the effects of 2 group exercises on functional status, quality of life and body composition and to show its correlation with sonographic measurements. There are 3 groups in total in the study. These are the control group given only the range of motion exercise, the second group given the range of motion and resistance exercise, and the third group given the range of motion and aerobic exercise. Exercise programs will last 12 weeks and it is planned to exercise 3 days a week.

DETAILED DESCRIPTION:
There are 3 groups in total in the study. The patients in the control arm will be given the practice of range of motion exercises for 50 minutes (1 day with a physiotherapist) 3 days a week for 12 weeks. The resistance exercise group will be given range of motion and resistance exercises with sandbag to the lower extremities for 12 weeks, 3 days a week for 50 minutes (1 day in the presence of a physiotherapist). In the aerobic exercise group, range of motion exercises and aerobic exercises on the treadmill will be given 50 minutes (1 day in the presence of a physiotherapist) 3 days a week for 12 weeks.

After the patient completes the 12-week exercise program, ultrasonographic measurements of transverse muscle thickness of M. Rectus femoris, vastus intermedius, long head of M.Biceps femoris and medial head of M. , 6-minute walk test, body composition measurements with DEXA device and quality of life measurements with SF-36, fatigue severity scale, fear assessment questionnaire in inflammatory rheumatic diseases and scales for other rheumatoid arthritis and pain status. Ultrasonographic measurements will be made at the midpoint between the anterior superior iliac spina and the upper end of the patella for rectus femoris and vastus intermedialis. For the medial head of the gascrokinemius, the measurement will be made at the thickest point where the head of the muscle is in the leg area, and for the biceps femoris muscle, 60% distal between the greater trochanter and the outer femoral condyle, and at the intersection point of a line drawn at the midline of the popliteal fossa. While measurements made for rectus femoris and vastus intermedius were evaluated in the supine position; The biceps femoris and gastrocnemius will be evaluated while the patient lies comfortably in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* Romatoid Arthritis diagnosed for> 1 year
* Female gender
* The patient has been in remission or low disease activity for at least 3 months
* 20-50 years

Exclusion Criteria:

* Patient with active arthritis or high disease activity
* Significant deformity and inability to ambulate in the lower extremity joints
* Pregnant patient
* Patient with menopause
* The presence of malignancy
* A patient with a serious psychiatric disorder and difficulty in cooperation
* Presence of cardiovascular and pulmonary comorbidity that may prevent exercise
* Male gender

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Muscle Size Measurement | at 12th week
  Ultrasonographic measurements of transverse muscle thickness will be made in M. Rectus femoris, vastus intermedius, long head of M. biceps femoris and medial head of M. Gastrocnemius. Ultrasonographic measurements will be made at the midpoint between the anterior superior iliac spina and the upper end of the patella for rectus femoris and vastus intermedialis. For the medial head of the gascrokinemius, the measurement will be made at the thickest point where the head of the muscle is in the leg area, and for the biceps femoris muscle, 60% distal between the greater trochanter and the outer femoral condyle and at the intersection point of a line drawn at the midline of the popliteal fossa. While measurements made for rectus femoris and vastus intermedius were evaluated in the supine position; The biceps femoris and gastrocnemius will be evaluated while the patient lies comfortably in the prone position.
5 chair test | at 12th week
  In the 5 chair test used in evaluating the functional status of the patient, "The practitioner allows the patient to sit on the chair with his back. The time it takes to sit and get up 5 times is measured with a stopwatch. " It will be made as.
Timed up and go test | at 12th week
  In the timed get up and walk test, "3 meters of space is determined in front of the patient sitting on a chair. The patient is asked to get up from the chair, walk this distance and sit down again. Elapsed time is measured with a stopwatch. " It will be applied as.
6-minute walking test | at 12th week
  In the 6-minute walking test, "The patient's goal should be to walk the longest distance that he can walk within 6 minutes. The longest distance that the patient can walk after 6 minutes is calculated in meters.
International Physical Activity Scale | at 12th week
  Those who score HIGH on the IPAQ engage in
  * Vigorous intensity activity on at least 3 days achieving a minimum total physical activity of at least 1500 MET minutes a week OR
  * 7 or more days of any combination of walking, moderate intensity or vigorous intensity activities achieving a minimum total physical activity of at least 3000 MET minutes a week.
  Scoring a MODERATE level of physical activity on the IPAQ means
  * 3 or more days of vigorous intensity activity and/or walking of at least 30 minutes per day OR
  * 5 or more days of moderate intensity activity and/or walking of at least 30 minutes per day OR
  * 5 or more days of any combination of walking, moderate intensity or vigorous intensity activities achieving a minimum total physical activity of at least 600 MET minutes a week.
  Scoring a LOW level of physical activity on the IPAQ means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.
Body Composition Measurements - Muscle | at 12th week
  In body composition measurements measured with the DEXA device, total muscle (kg) and their ratio to the total body will be calculated.
Body Composition Measurements - Fat | at 12th week
  In body composition measurements measured with the DEXA device, total fat mass according to regions (kg) and their ratio to the total body will be calculated.
Body Composition Measurements - Soft tissue | at 12th week
  In body composition measurements measured with the DEXA device, total soft tissue mass (kg) and their ratio to the total body will be calculated.
Short Form - 36 | at 12th week
  In the evaluation with the short form-36, it is aimed to learn the patient's views about her own health, how she feels and how much she can perform her daily activities. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Visual Pain Scale | at 12th week
  Visual pain scale scored from 0 (no pain) to 10 (maximal pain) will be used in the global pain assessment of the patient.
Fear assessment questionnaire in inflammatory rheumatic diseases | at 12th week
  Fear assessment questionnaire in inflammatory rheumatic diseases will be filled. Minimum value is 0, maximum value is 100. Higher score is worse result
Body mass index | at 12th week
  Body mass index (weight and height will be combined to report BMI in kg/m^2) will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayyildiz A, Yilmaz F, Altindas H, Ciftci S, Kuran B. Effects of Aerobic and Resistive Exercise on Muscle Measurements and Body Composition in Female Patients With Rheumatoid Arthritis. Am J Phys Med Rehabil. 2023 Dec 1;102(12):1076-1084. doi: 10.1097/PHM.0000000000002283. Epub 2023 May 10. PMID 37204935